CLINICAL TRIAL: NCT07005739
Title: Effectiveness of Turkish Folk Dance Exercises on Core Stabilization, Balance, and Agility in U14 Football Players
Brief Title: Turkish Folk Dance Exercises in Core Stabilization, Balance, and Agility Training for U14 Football Players
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2022.386
Record Dates: First submitted 2025-05-26; First posted 2025-06-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Physical Performance Enhancement; Motor Skills Development; Agility, Balance, and Core Stabilization in Youth Athletes
Keywords: Folk dances,; Kinesthetic sense; Core region stability; Youth football; Balance; Turkish folk dance; Agility; core stability; flexibility; proprioception; exercise intervention; sports performance; U14 athletes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Folk Dance + Football Training Group: Participants (n=15) who received Turkish folk dance-based exercises in addition to regular football training for 8 weeks.
  Interventions: Behavioral: Turkish Folk Dance-Based Exercise Program
- Football-Only Training Group: Participants (n=15) who continued only their regular football training for 8 weeks.

INTERVENTIONS:
Behavioral: Turkish Folk Dance-Based Exercise Program — Participants in the intervention group received a structured Turkish folk dance-based exercise program in addition to their regular football training. The dance-based intervention consisted of two 45-minute sessions per week for 8 weeks, including traditional Turkish folk dance movements aimed at improving balance, agility, and core stability.
  Groups: Folk Dance + Football Training Group

SUMMARY:
This study aims to examine the effects of integrating Turkish folk dance exercises into the training routines of U14 football players on their kinesthetic sense, balance, agility, core stabilization, and flexibility. The study includes 15 young male football players actively participating in league matches in Istanbul, randomly assigned to either control or intervention groups. The intervention group participates in an additional Turkish folk dance training program for eight weeks alongside their regular football practice, while the control group continues with regular training only. Both groups undergo assessments on agility, flexibility, core stabilization, balance, and kinesthetic sense using standardized field tests. The study seeks to explore whether Turkish folk dance training can provide added value to conventional youth football training programs.

DETAILED DESCRIPTION:
This randomized controlled study investigates the potential impact of Turkish folk dance-based exercises on core region stabilization, balance, and agility among U14 male football players in Istanbul. Fifteen participants are divided into control and experimental groups. The experimental group participates in an eight-week Turkish folk dance exercise program in addition to their regular football training. Pre- and post-intervention assessments include the Illinois Agility Test, Y-Balance Test, joint position sense measurements, flexibility assessments, and the Core Stabilization Test (CST). Statistical analysis methods planned for evaluating the outcomes include normality analysis, independent samples t-tests for group comparisons, and paired samples t-tests for within-group differences, with a significance level set at p<0.05. The study aims to assess whether incorporating Turkish folk dance movements into youth football training programs may contribute to improvements in motor skills relevant to athletic performance and injury prevention.

ELIGIBILITY:
Inclusion Criteria:

* Male football players actively participating in the U14 league in Istanbul.
* Age between 12 and 14 years.
* Actively training and participating in official football matches.
* Voluntary participation with parental/guardian consent.

Exclusion Criteria:

* Presence of musculoskeletal, neurological, or chronic health conditions that would prevent participation.
* History of injury or surgery affecting balance or mobility within the last 6 -months.
* Participation in other structured exercise or dance programs outside of football training.
* Non-compliance with the training or assessment schedule.

Ages: 12 Years to 14 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Male U14 football players actively competing in the Istanbul youth football league. Participants were healthy, regularly training, and had no existing injuries or chronic health conditions affecting physical performance.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Agility Performance | Baseline and post-intervention (8 weeks)
  Change in agility measured by the Illinois Agility Test, assessed before and after the 8-week intervention period.
Balance Performance | Baseline and post-intervention (8 weeks)
  Change in dynamic balance measured by the Y-Balance Test, assessed before and after the 8-week intervention period.
Core Stabilization | Baseline and post-intervention (8 weeks)
  Change in core stabilization measured by the Core Stabilization Test (CST), assessed before and after the 8-week intervention period.

SECONDARY OUTCOMES:
Flexibility | Baseline and post-intervention (8 weeks)
  Change in flexibility assessed by the Passive Straight Leg Raise Test, before and after the intervention.
Kinesthetic Sense / Joint Position Sense | Baseline and post-intervention (8 weeks)
  Change in kinesthetic sense measured by Joint Position Sense (JPS) testing, before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tuba KIZILET TOPATEŞ, Prof., Study Director — Marmara University, Faculty of Sport Sciences, Istanbul, Turkey; Ceren AĞAOĞLU TOPÇU, Dr., Principal Investigator — Marmara University, Faculty of Sport Sciences, Istanbul, Turkey
Locations (2):
- Turkey (Türkiye) (2):
  - Başakşehir Spor Kulübü, Istanbul, Başakşehir
  - Yakuplu Spor Kulübü, Istanbul, Beylikdüzü

IPD SHARING:
Plan to Share IPD: No
The study protocol does not include provisions for sharing individual participant data (IPD) outside the research team, in accordance with participant privacy and institutional regulations.